CLINICAL TRIAL: NCT03387319
Title: Social Stress, Inflammation, and Chronic Kidney Disease Among African Americans
Brief Title: Stress and CKD Among African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kimberly R Jacob Arriola, PhD, MPH, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00099892; 1R21DK112108 (NIH)
Record Dates: First submitted 2017-12-20; First posted 2018-01-02 (Actual); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Chronic Kidney Disease
Keywords: Social stress; Inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation

STUDY DESIGN:
Intervention Model Description: Of the 100 participants recruited, 80 will have a diagnosis of chronic kidney disease (CKD) and 20 will not. Participants will be randomized such that half will recall the racial experience and half will recall the non-racialized stressful event. Each participant will have an equal chance of being placed in the racialized or non-racialized experience group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Racialized Stressful Event Recall (Experimental): Participants in this study are recall a stressful event related to race.
  Interventions: Behavioral: Racialized Stressful Event Recall
- Non-racialized Stressful Event Recall (Experimental): Participants in this study arm recall a stressful event unrelated to race.
  Interventions: Behavioral: Non-Racialized Stressful Event Recall

INTERVENTIONS:
Behavioral: Racialized Stressful Event Recall — Participants will undergo a moderate psychological stress adapted from the Trier Social Stress Test (TSST) where they will be asked to recall a stressful, real-life, race-related event.
  After instructions are provided, participants will be given two minutes to prepare their statement, and three minutes to deliver their statement. There will be an 'audience' present at each participant's speaking task which will include two observers who are of same race as the participant (African American), to heighten stress responses.
  Arms: Racialized Stressful Event Recall
Behavioral: Non-Racialized Stressful Event Recall — Participants will undergo a moderate psychological stress adapted from the Trier Social Stress Test (TSST) where they will be asked to recall a stressful, real-life, event unrelated to race.
  After instructions are provided, participants will be given two minutes to prepare their statement, and three minutes to deliver their statement. There will be an 'audience' present at each participant's speaking task which will include two observers who are of same race as the participant (African American), to heighten stress responses.
  Arms: Non-racialized Stressful Event Recall

SUMMARY:
The goal of this study is to determine whether experiencing stress from discrimination may increase chronic kidney disease (CKD) progression in African Americans. Study participation occurs over the course of 2 days, and participant time burden is expected to be about 4.5 hours, plus a 24-hour period of wearing a blood pressure monitor.

DETAILED DESCRIPTION:
On Day 1, the project coordinator will explain the study to participants and answer any questions he/she may have. Those who agree to participate in the study will provide consent at the clinic and will also be asked to complete a questionnaire on an iPad in a small, private room at the clinic. The participant will complete the questionnaire alone, however, the project coordinator will read questions aloud if the participant chooses. Before leaving on Day 1, participants will fitted with a blood pressure monitor to be worn for the next 24 hours.

The clinical intervention portion of the study occurs during the morning of Day 2 (between 9:00 AM and 11:00 AM). Participants will be instructed to bring the blood pressure monitor and a list of current medications (or the actual medications) with them. First, participants will provide a urine sample and undergo blood pressure testing. A research nurse will insert a catheter (a small thin tube) into the participant's vein, and allow a 30-minute resting period so that the participant gets used to the catheter, and then take a baseline blood draw. Participants will judge how distressed they feel in that moment using a standard scale and tell the project coordinator his/her rating. Next, participants will be randomized to one of two study arms such that half will recall the racial experience and half will recall the non-racialized stressful event. An audience of two observers of same race will wear white coats and watch as the participants recall the stressful events. The research nurse will draw blood and take blood pressure measurements at multiple time points during both recall experiences. Immediately before and after each recall task, the participant will again judge how distressed he/she is feeling in that moment using the same scale as before. The project coordinator will explain the purpose of the story recall and common ways that individuals may respond to the task (such as feeling anxious after the task). A total of 100 people will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Emory University Hospital Midtown
* Self-identify as African American or Black
* Estimated glomerular filtration rate (eGFR) ≥ 15, or <90

Exclusion Criteria:

* Mental disorder that prevents the completion of the Computer Assisted Personal Interview (CAPI) and the stressful recall manipulation
* Currently on maintenance dialysis
* Unable or unwilling to undergo intravenous catheterization

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Arriola, PhD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arriola KJ, Lewis TT, Pearce B, Cobb J, Weldon B, Valentin MIZ, Lea J, Vaccarino V. A randomized trial of race-related stress among African Americans with chronic kidney disease. Psychoneuroendocrinology. 2021 Sep;131:105339. doi: 10.1016/j.psyneuen.2021.105339. Epub 2021 Jun 18. PMID 34175554

RESULTS

PARTICIPANT FLOW:
Groups:
- Racialized Stressful Event Recall: Participants in this study arm recalled a stressful event related to race.
- Non-racialized Stressful Event Recall: Participants in this study arm recalled a stressful event unrelated to race.
Period: Overall Study
Arm/Group | Racialized Stressful Event Recall | Non-racialized Stressful Event Recall
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Racialized Stressful Event Recall | Non-racialized Stressful Event Recall | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.92 (8.66) | 50.12 (9.57) | 52.52 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 9 | 11 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 25 | 50
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Subjective Units of Distress Scale (SUDS) Score
Description: Level of distress will be measured with the Subjective Units of Distress Scale (SUDS). Participants rate their distress on a linear scale from 0 to 100, where 0 = No distress; totally relaxed, 50 = Moderate anxiety/distress; uncomfortable, but can continue to function, 100 = Highest anxiety/distress ever felt. The SUDS will be administered at baseline and after the first stress task. The change in SUDS scores is presented here. Scores above zero mean that the participants experienced an increase in distress following the stress task.
Time Frame: Baseline (Minute 0), Minute 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Racialized Stressful Event Recall | Non-racialized Stressful Event Recall
Number analyzed (Participants) | 25 | 25
score on a scale | 2.92 (2.74) | 3.12 (3.07)

2. Primary Outcome: Change in Cooper's Racism Recall Scale Score
Description: Participants will report their level of stress directly related to reliving the stressful experience using an adapted version of Cooper's Racism Recall Scale. Participants reported their level of distress at the time of the event and currently while thinking about the event, on a linear scale from 0 to 10 where higher values indicate higher distress. Values presented here are the change from baseline and values greater than 0 mean that stress increased from before (baseline) and after the stressful event recall.
Time Frame: Baseline (Minute 0), Minute 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Racialized Stressful Event Recall | Non-racialized Stressful Event Recall
Number analyzed (Participants) | 25 | 25
score on a scale | 6.24 (2.57) | 5.48 (3.57)

3. Primary Outcome: Change in Monocyte Chemoattractant Protein-1 (MCP-1) Level
Description: Monocyte Chemoattractant Protein-1 (MCP-1) is an inflammatory marker that is sensitive to acute stress induction and is associated with chronic kidney disease (CKD). Blood will be drawn three times, at 30 minutes after the IV catheter is inserted (prior to the stressful event recall) and after each 45 minute recovery period following the stress tests, in order to compare MCP-1 levels at before and after the study intervention. Increased MCP-1 indicates an increased inflammatory response. MCP-1 levels will be quantitated by the MesoScale system (MSD Rockville, Maryland) according to the protocols supplied by the manufacturer, which uses electrochemiluminescence for high sensitivity with a dynamic range of 0.09-375 pg/mL. Values presented here are the difference between the baseline and post-intervention blood draws and values greater than 0 indicate that there is an increase in inflammatory response post-intervention.
Time Frame: Baseline (Minute 0), Minute 90 (after both stress tests and rest periods)
Population: Lab values are missing for 15 participants due to lab error.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Racialized Stressful Event Recall | Non-racialized Stressful Event Recall
Number analyzed (Participants) | 18 | 17
pg/mL | 193.12 (92.80) | 217.31 (110.47)

4. Primary Outcome: Change in Interleukin-6 (IL-6) Level
Description: Interleukin-6 (IL-6) is an inflammatory marker that is sensitive to acute stress induction and is associated with CKD. Blood will be drawn three times, at 30 minutes after the IV catheter is inserted (prior to the intervention) and after each 45 minute recovery period following the stress tests, in order to compare IL-6 levels at before and after the study intervention. IL-6 is influenced by a variety of factors and increases in IL-6 indicate an increased inflammatory response. IL-6 levels will be quantitated by the MesoScale system (MSD Rockville, Maryland) according to the protocols supplied by the manufacturer, which uses electrochemiluminescence for high sensitivity with a dynamic range of 0.06-488 pg/mL. Values presented here are the difference between the baseline and post-intervention blood draws and values greater than 0 indicate that there is an increase in inflammatory response post-intervention.
Time Frame: Baseline (Minute 0), Minute 90 (after both stress tests and rest periods)
Population: Lab values are missing for 15 participants due to lab error.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Racialized Stressful Event Recall | Non-racialized Stressful Event Recall
Number analyzed (Participants) | 18 | 17
pg/mL | 2.23 (1.02) | 2.11 (1.29)

5. Primary Outcome: Change in Soluble Urokinase-type Plasminogen Activator Receptor (suPAR) Level
Description: Soluble urokinase-type plasminogen activator receptor (suPAR) is an inflammatory marker that is sensitive to acute stress induction and is associated with CKD. Blood will be drawn three times at 30 minutes after the IV catheter is inserted (prior to the intervention) and after each 45 minute recovery period following the stress tests, in order to compare suPAR levels at before and after the study intervention. Increases in suPAR indicate an increased inflammatory response. suPAR will be measured with the Virogates (CEDARLANE Laboratories, Burlington, NC) suPARnostic® ELISA, according to the protocols supplied by the manufacturer. This assay has a high sensitivity (0.1 ng/mL) giving consistently quantitative results in plasma samples. Values presented here are the difference between the baseline and post-intervention blood draws and values greater than 0 indicate that there is an increase in inflammatory response post-intervention.
Time Frame: Baseline (Minute 0), Minute 90 (after both stress tests and rest periods)
Population: Lab values are missing for 15 participants due to lab error.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Racialized Stressful Event Recall | Non-racialized Stressful Event Recall
Number analyzed (Participants) | 18 | 17
ng/mL | 4.18 (1.66) | 4.50 (1.50)

6. Primary Outcome: Change in Systolic Blood Pressure
Description: Blood pressure readings will be taken at baseline and every 5 minutes during the experimental manipulation, except during the recall task when blood pressure will be measured every 1 minute. Mean systolic blood pressure scores for rest, recall task, and recovery will be calculated by averaging the readings taken during each period. Blood pressure reactivity will be a change score, calculated as the mean of the scores during the recall task minus the mean of the scores during rest, designed to represent the change in systolic blood pressure induced by the recall task. Values greater than 0 are the mean increase in systolic blood pressure following the intervention, compared to the baseline time period.
Time Frame: Prior to IV insertion at Minute -30 through Minute 130
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Racialized Stressful Event Recall | Non-racialized Stressful Event Recall
Number analyzed (Participants) | 25 | 25
millimeters of mercury (mmHg) | 11.79 (12.76) | 15.72 (19.20)

7. Primary Outcome: Change in Diastolic Blood Pressure
Description: Blood pressure readings will be taken at baseline and every 5 minutes during the experimental manipulation, except during the recall task when blood pressure will be measured every 1 minute. Mean diastolic blood pressure scores for rest, recall task, and recovery will be calculated by averaging the readings taken during each period. Blood pressure reactivity will be a change score, calculated as the mean of the scores during the recall task minus the mean of the scores during rest, designed to represent the change in diastolic blood pressure induced by the recall task. Values greater than 0 are the mean increase in diastolic blood pressure following the intervention, compared to the baseline time period.
Time Frame: Prior to IV insertion at Minute -30 through Minute 130
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Racialized Stressful Event Recall | Non-racialized Stressful Event Recall
Number analyzed (Participants) | 25 | 25
millimeters of mercury (mmHg) | 5.52 (6.15) | 7.59 (8.37)

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from the time the participant consents to take part in the study (Day 1) through the experimental manipulation on Day 2.
Arm/Group | Racialized Stressful Event Recall | Non-racialized Stressful Event Recall
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT03387319/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT03387319/ICF_001.pdf